CLINICAL TRIAL: NCT06206889
Title: Nursing Activity Score (Nursing Activities Score-NAS) Verification of Turkish Version
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Ozgur Komurcu, principle investigator intensivist, Samsun University
Other Study IDs: SUKAEK 2023-12/2
Record Dates: First submitted 2023-12-20; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Nurse's Role
Keywords: validation; NAS
MeSH Terms: interventions — nas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nurse: Nurses working in tertiary intensive care
  Interventions: Other: NAS

INTERVENTIONS:
Other: NAS — NAS Turkish language validation will be carried out. NAS and CNSI scores will be recorded during the shifts of nurses serving patients in Level 3 intensive care units by the nurse in charge and another independent evaluator, and the correlation between the two scores will be investigated.
  Other Names: CNSI

SUMMARY:
Various tools for measuring nursing workload have been described in the national and international literature. For this purpose, Cullen et al. The Therapeutic Intervention Scoring System (TISS)-28, created by Miranda et al. Nursing Activities Score (NAS) was created by revising by. NAS covers 80.8% of all nursing activities, surpassing the 43.3% coverage of TISS-28.

Critical Nursing Situation Index (CNSI) has been validated and adapted in our country and has been found to be a valid and reliable scale for the Turkish society. The aim of this study is to adapt the Nursing Activities Score (NAS) to Turkish and determine its correlation with CNSI scores.

DETAILED DESCRIPTION:
Various tools for measuring nursing workload have been described in the national and international literature. The Therapeutic Intervention Scoring System (TISS)-28, which is designed to classify the nursing workload of patients in intensive care units according to the severity of their illness to be evaluated by a panel of experts, evaluates 43.3% of nursing activities. Miranda et al. In order to reduce possible erroneous evaluations, some changes were made to TISS-28 and the Nursing Activities Score (NAS) was created. NAS covers 80.8% of all nursing activities, surpassing the 43.3% coverage of TISS-28.

The Critical Nursing Situation Index (CNSI), which was finalized with 84 items developed by Binnekade et al., was validated and adapted in our country and was found to be a valid and reliable scale for the Turkish society.

In this study, which was carried out to adapt and validate the Nursing Activities Score (NAS) into Turkish, the internal consistency Cronbach's alpha coefficient was found to be p = 0.718 after a pilot study with a sample of 30 adult intensive care patients and 30 nurses. After the significant internal consistency obtained in the pilot study, it was aimed to examine the correlation of NAS internal consistency and CNSI scores in 150 work shift.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who serve patients over the age of 18 who stay in Level 3 intensive care for at least 24 hours

Exclusion Criteria:

* Those nurses; Serving patients under the age of 18, Caring for patients who are scheduled to be discharged from intensive care within 24 hours, Those who change their workplace for any reason during the work shift Who did not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses providing 3rd level intensive care services at Samsun University
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of NAS Turkish validity and applicability | 6 month
  NAS was developed to measure the workload of nurses in patient care. Scores refer to the average time spent caring for patients, not the severity of the disease. Total NAS can range from 0 to 177 points. A score above 100 points indicates that more than one nurse is needed to provide care.

SECONDARY OUTCOMES:
Investigating the correlation between NAS and CNSI | 6 month
  CNSI, which has previously been validated in Turkish, will be applied together with NAS in the same nurse shift, so that the correlation between the two scores will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Özgür Kömürcü, Study Director — Samsun University
Locations (1):
- Özgür Kömürcü, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Binnekade JM, de Mol BA, Kesecioglu J, de Haan RJ. The Critical Nursing Situation Index for safety assessment in intensive care. Intensive Care Med. 2001 Jun;27(6):1022-8. doi: 10.1007/s001340100947. PMID 11497134
- [Background] Cullen DJ, Civetta JM, Briggs BA, Ferrara LC. Therapeutic intervention scoring system: a method for quantitative comparison of patient care. Crit Care Med. 1974 Mar-Apr;2(2):57-60. No abstract available. PMID 4832281
- [Background] Miranda DR, Nap R, de Rijk A, Schaufeli W, Iapichino G; TISS Working Group. Therapeutic Intervention Scoring System. Nursing activities score. Crit Care Med. 2003 Feb;31(2):374-82. doi: 10.1097/01.CCM.0000045567.78801.CC. PMID 12576939